CLINICAL TRIAL: NCT01267643
Title: A Phase 1/2 Study of Alefacept, a CD2 Receptor Antagonist in Patients With Relapsed/Refractory Aplastic Anemia
Brief Title: Alefacept in Patients With Relapsed/Refractory Aplastic Anemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug not available at this time
Sponsor: The Cleveland Clinic (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5Z10; CASE 5Z10 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-12-20; First posted 2010-12-28 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Aplastic Anemia
Keywords: Alefacept; Amevive; Aplastic Anemia; Moderate to Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alefacept (Experimental)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — Dose Escalation Schedule
  Level -1 5 mg IV once weekly
  Level 1 7.5 mg IV once weekly
  Level 2 10 mg IV once weekly
  Level 3 12.5 mg IV once weekly
  Other Names: Amevieve

SUMMARY:
Aplastic Anemia (AA) is an autoimmune hematologic stem cell disease mediated by activated T-lymphocytes that leads to pancytopenia. The disease related morbidity and mortality if left untreated can approach 90%. For over 30 years, anti-thymocyte globulin (ATG) in combination with cyclosporine (CsA) remains the standard therapy. However, the treatment response with ATG is at best between 50-60% with a sizeable number of partial responses. Treatment with ATG is also associated with significant toxicity and high relapse rate that can be as high as 45%. Since the prognosis in refractory and relapsed AA remains poor, there is a need for less toxic novel immunosuppressive agents that can improve response rates and remission duration in refractory and relapsed AA.

Alefacept is a human recombinant dimeric fusion protein composed of the terminal portion of leukocyte functioning antigen-3 (LFA3/CD58) and the Fc portion of human IgG1. It prevents co-stimulatory signals between antigen presenting cells and memory T cells by competitive inhibition of CD2 in T cells, induces selective apoptosis of CD4+ and CD8+ memory effector T cells by interaction between the Fc portion of IgG1 and the FcyIII in NK cells, and possibly direct ligation of CD2 molecules on T cells that subsequently result in the alteration in T cell agonist signaling. It has been used successfully in the treatment of other T cell mediated disorders particularly psoriasis and steroid refractory graft versus host disease (GVHD) with minimal side effects. In a case of liver transplant associated AA (similar to transfusion associated AA) which is fatal in most patients, Alefacept induced remission after patient did not respond to ATG and other immunosuppressants. The investigators hypothesize that the LFA3-CD2 co-stimulatory pathway play an important role in the immune pathogenesis of AA and treatment with Alefacept can help treat refractory/relapsed cases of AA.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Primary Objective

   * To define the safety, tolerability, dose-limiting toxicities (DLT), of alefacept in relapsed/ refractory aplastic anemia (AA).
   * To evaluate the efficacy of alefacept in refractory/ relapsed AA by determining overall response rates (ORR) which includes complete remission [CR] and partial remission (PR) rates.
2. Secondary Objective

   * To evaluate for predictive markers for response to Alefacept with relapsed/ refractory AA and evaluate its effect on the PNH clone. The effects of alefacept in major populations of lymphocytes will be evaluated. The absolute numbers of various T cell populations including CD3+ T cell, CD3+/CD4+ T cell, CD3+/CD8+, CD57+ natural killer cell count and CD4/CD8 ratio will be measured as part of an immunodeficiency panel by flow cytometry. The functional properties of T cells will be evaluated by measuring markers of T cell activation and cytokine production. The saturation of CD2 receptors with alefacept will be determined. Occupied CD2 will not be detectable by competing antibody in-vitro. The expression of CD2 within lymphocytes will be measured prior to the initiation of therapy and every 2 weeks prior to and 30 minutes after the administration of alefacept. The presence of a Paroxysmal Nocturnal Hemoglobinuria (PNH) clone in patients with AA has been shown to correlate with increased response to immunosuppression25.

OUTLINE: This is an open-label, single center study. Patients will receive intravenous Alefacept once weekly for a total of 12 weeks in the absence of disease progression or unacceptable toxicity. After completion of the 12 week treatment, patients will go through a 12 week observation period. After completion of the study, patients will be followed periodically. The dose defined in the Phase 1 study will be used for the subsequent Phase 2 study. Four bone marrow biopsies will be taken at screening, week 13, week 24, and the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilled criteria for diagnosis of either moderate (mAA) or severe aplastic anemia (sAA) at the time of initial diagnosis defined per protocol.
2. Patient with a history sAA must have had an incomplete response at least 3 months following treatment with ATG/CsA, or they must have relapsed following an initial response to treatment.
3. Patient must not be receiving any cyclosporine or any other T cell immunosuppressive agents within 4 weeks of study entry.
4. Patients must have organ function as defined below:

   * total bilirubin within normal institutional limits (NV: 0.0-1.5 mg/dL)
   * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal AST (NV: 7-40 U/L); ALT (NV: Male 5-50 U/L; Female 0-45 U/L)
   * creatinine within normal institutional limits (NV: Age 18 0.4-1.3 mg/dL; 19-99 years old 0.7-1.4 mg/dL) OR
   * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
5. Peripheral blood counts at the time of enrollment must include at least one of the following: Hgb <9 g/dL or red blood cell (RBC) transfusion dependence, ANC <1000/µl, or platelet count of <60,000/µL.
6. Women of child-bearing potential and men must agree to use adequate contraception defined per protocol.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents (other than hematopoietic growth factors) within 4 weeks of study entry.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Alefacept.
3. Current diagnosis of acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), Fanconi's anemia, Dyskeratosis Congenita (DC) or other hereditary forms of AA.
4. Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent.
5. Age <18 years.
6. ECOG performance status >2 (Karnofsky <60%, see Appendix A).
7. Malignancy other than non-melanoma skin cancer within the last 2 years.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined as uncontrolled infection requiring IV antibiotics, invasive fungal infection and progressive CMV viremia), symptomatic congestive heart failure (NYH class III and IV), unstable angina pectoris, or cardiac arrhythmia.
9. Pregnant or breastfeeding women.
10. HIV-positive patients on combination antiretroviral therapy.
11. Patients who have previously received systemic chemotherapy and/ or radiation therapy.
12. Patients who previously underwent allogeneic hematopoietic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12-16 (Actual); Study Completion 2013-04-16 (Actual)

PRIMARY OUTCOMES:
To measure the number of dose limiting toxicities (DLTs) as a determination of the maximum tolerable dose (MTD). | Every 12 weeks
  The dosing cohorts includes (Cohort -1= 5 mg IV weekly, Cohort 1= 7.5 mg IV weekly, Cohort 2= 10 mg IV weekly, and Cohort 3= 12.5 mg IV weekly). The MTD will be defined as the dose level that has maxiumum effectiveness with minimal toxicity.
To evaluate the efficacy of alefacept in refractory/ relapsed AA by determining overall response rates (ORR) which includes complete remission [CR] and partial remission (PR) rates. | Every 12 weeks

SECONDARY OUTCOMES:
To analyze bood samples to evaluate for predictive markers for response to Alefacept with relapsed/ refractory AA and evaluate its effect on the PNH clone. | Every 2 weeks for the first 4 weeks, then monthly after that

CONTACTS AND LOCATIONS:
Overall Officials: Ramon V. Tiu, M.D., Principal Investigator — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States